CLINICAL TRIAL: NCT07013019
Title: Reference Values for Knee Rotational Amplitudes in a Population of Athletes
Acronym: PRELAX
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-CHITS-008
Record Dates: First submitted 2025-05-27; First posted 2025-06-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Knee Ligament Injury
Keywords: Anterior cruciate ligament; Injury; Laxity; Pivot sport; Dynamic arthrometer
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy male and female athletes aged 15 and over practising competitive pivot sports
  Interventions: Other: Measures of overall (internal+external) knee rotational amplitudes

INTERVENTIONS:
Other: Measures of overall (internal+external) knee rotational amplitudes — Measures of overall (internal+external) knee rotational amplitudes by Dyneelax

SUMMARY:
Rupture of the anterior cruciate ligament (ACL) is a frequent and disabling injury in pivot sports, leading to knee laxity and instability, reduced performance and an increased risk of early osteoarthritis. The risk is 2 to 8 times higher in women, linked to greater ligament laxity and a different quadriceps/hamstring muscle ratio post-puberty.

To assess knee laxity and the degree of ligament damage, anterior tibial translation (of the tibia below the femur) is usually measured. This translation is symmetrical and varies between 3 and 10 mm depending on the individual (natural laxity). It is increased in cases of ACL damage.

Measuring tibial rotation is also of interest in this context. Studies show that the ACL plays a crucial role in controlling internal and external tibial rotation, especially during low-flexion movements (between 10° and 30°). ACL rupture also significantly increases this rotation, aggravating knee instability.

It therefore seems important to study both tibial rotation and tibial translation to assess knee laxity. Combining these two measurements seems to improve diagnostic accuracy. This multifactorial approach could provide additional information on biomechanical abnormalities and predisposition to injury. The use of biomechanical data, such as normative values for tibial rotation, is fundamental to prevention, and preventive exercise programs reduce the risk of rupture4. Defining these norms would help identify athletes at risk and personalize preventive strategies.

Instrumented assessment of laxity, using devices such as the DYNEELAX dynamic arthrometer, enables precise quantification of tibial rotation and anterior tibial translation under controlled loads. Its reliability has been proven5 and its use has been mastered at Toulon ("Unité de Médicine et Traumatologie du Sport") and Brest (Centre de Médecine du Sport"). It will be used in the PRELAX project to define normative tibial rotation values.

DETAILED DESCRIPTION:
This retrospective and prospective multicenter observational study aims to define normative values for overall (internal+external) knee rotational amplitudes in a population of healthy male and female athletes aged 15 and over, practising competitive pivot sports (between 2022 and 2026). Data will be collected in 2 centers: Toulon ("Unité de Médicine et Traumatologie du Sport") and Brest (Centre de Médecine du Sport").

ELIGIBILITY:
Inclusion Criteria:

1. Athletes with healthy knees, men and women ;
2. Age greater than or equal to 15 years;
3. Competitive pivot sports.

Exclusion Criteria:

1. History of ligament, meniscus, cartilage or bone lesions in the knee ;
2. Pain, stiffness or instability in the knee at the time of inclusion;
3. Knee surgery, including ligament reconstruction;
4. Systemic diseases or medical conditions that may affect the musculoskeletal system;
5. Opposition of the participant and/or his/her legal representative in the case of a minor participant;
6. Participant under protective supervision.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy male and female athletes aged 15 and over practising competitive pivot sports and consulted at Toulon ("Unité de Médicine et Traumatologie du Sport") and Brest (Centre de Médecine du Sport") as part of their sports medicine follow-up
Sampling Method: Non-Probability Sample
Enrollment: 482 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Measures of overall (internal+external) knee rotational amplitudes | day of medical examination (day 1)
  Values of maximum knee rotational amplitudes (internal and external) measured by the DYNEELAX arthrometer: maximum internal and maximum external tibial rotation in degrees, taking into account the overall amplitude.

SECONDARY OUTCOMES:
Global rotation asymmetries between the two knees | day of medical examination (day 1)
  Percentage of participants with significant asymmetry between left and right knees and level of asymmetry by calculating the mean and standard deviation of the asymmetry index
Correlation between rotational and translational laxity | day of medical examination (day 1)
  Assessment of the strength and direction of the correlation between rotational and translational laxity with a Pearson correlation coefficient (varies between 0 and 1)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques Raymond, MD, Study Director — Centre Hospitalier Intercommunal Toulon La Seyne sur Mer; Christophe GUEGAN, MD, Principal Investigator — Centre de Médecine du Sport de Brest
Locations (2):
- France (2):
  - Centre Hospitalier Intercommunal Toulon La Seyne sur Mer, Toulon, Var
  - Centre de Médecine du Sport, Brest

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmad CS, Clark AM, Heilmann N, Schoeb JS, Gardner TR, Levine WN. Effect of gender and maturity on quadriceps-to-hamstring strength ratio and anterior cruciate ligament laxity. Am J Sports Med. 2006 Mar;34(3):370-4. doi: 10.1177/0363546505280426. Epub 2005 Oct 6. PMID 16210574
- [Background] Andersen HN, Dyhre-Poulsen P. The anterior cruciate ligament does play a role in controlling axial rotation in the knee. Knee Surg Sports Traumatol Arthrosc. 1997;5(3):145-9. doi: 10.1007/s001670050042. PMID 9335025
- [Background] Mouton C, Theisen D, Meyer T, Agostinis H, Nuhrenborger C, Pape D, Seil R. Combined anterior and rotational knee laxity measurements improve the diagnosis of anterior cruciate ligament injuries. Knee Surg Sports Traumatol Arthrosc. 2015 Oct;23(10):2859-67. doi: 10.1007/s00167-015-3757-7. Epub 2015 Aug 30. PMID 26318487
- [Background] Arundale AJH, Bizzini M, Dix C, Giordano A, Kelly R, Logerstedt DS, Mandelbaum B, Scalzitti DA, Silvers-Granelli H, Snyder-Mackler L. Exercise-Based Knee and Anterior Cruciate Ligament Injury Prevention. J Orthop Sports Phys Ther. 2023 Jan;53(1):CPG1-CPG34. doi: 10.2519/jospt.2023.0301. PMID 36587265
- See also: Cojean T, Batailler C, Robert H, Cheze L. Sensitivity, repeatability and reproducibility study with a leg prototype of a recently developed knee arthrometer: The DYNEELAX®. Med Nov Technol Devices. 2023 Sep 1. doi: 10.1016/j.medntd.2023.100254 — https://doi.org/10.1016/j.medntd.2023.100254